CLINICAL TRIAL: NCT07357831
Title: A Randomized, Multicenter, Investigator-Blind Phase III Trial To Evaluate The Efficacy And Safety Of MC2-01 Cream Compared To CAL/BDP Gel and Vehicle In Chinese Subjects With Plaque Psoriasis
Brief Title: A Phase III Trial To Evaluate The Efficacy And Safety Of MC2-01 Cream Compared To CAL/BDP Gel and Vehicle In Plaque Psoriasis Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Collaborators: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDM3015-301
Record Dates: First submitted 2025-12-11; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MC2-01 Cream (Experimental): MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream. One application daily for 8 weeks
  Interventions: Drug: MC2-01 cream
- MC2-01 Vehicle (Sham Comparator): One application daily for 8 weeks.
  Interventions: Drug: MC2-01 vehicle
- CAL/BDP Gel (Active Comparator): Calcipotriene/betamethasone (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%). One application daily for 8 weeks.
  Interventions: Drug: CAL/BDP Gel

INTERVENTIONS:
Drug: MC2-01 cream — MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  Arms: MC2-01 Cream
Drug: MC2-01 vehicle — Vehicle Cream
  Arms: MC2-01 Vehicle
Drug: CAL/BDP Gel — calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%
  Arms: CAL/BDP Gel

SUMMARY:
This is a multi-center, randomized, investigator-blinded, calcipotriol and betamethasone dipropionate gel and vehicle-controlled phase 3 clinical study to evaluate the efficacy and safety of MC2-01 cream in the treatment of Chinese plaque psoriasis to assess the efficacy and safety of MC2-01 cream in Chinese subjects aged ≥ 18 years with plaque psoriasis. This study includes a screening period, a treatment period, and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the objectives and requirements of this study, voluntarily participate in the clinical trial and sign the informed consent form (ICF), and be able to complete all visits as required by the protocol.
2. Aged ≥ 18 years at the time of signing the ICF, male or female.
3. Clinical diagnosis of plaque psoriasis with involvement of the body (trunk and/or limbs) before the first dose of this study, with a disease duration of ≥ 6 months and stable for the last 4 weeks.
4. Subjects are required to meet the following requirements at screening and baseline:

   * BSA of psoriatic involvement on body (trunk and/or limbs) ranging from 2% to 30%, with total BSA not exceeding 30% if scalp involvement is present;
   * Body (trunk and/or limbs) PGA score of 2 or 3;
   * mPASI score ≥3.
5. Female of childbearing potential (WOCBP) subjects with a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline. WOCBP and male subjects who have not received a vasectomy must agree to take at least one effective method of contraception, including oral/implantable/injectable/transdermal contraceptive, intrauterine device, bilateral tubal ligation or occlusion, vasectomy, and barrier contraception (used correctly and throughout sexual intercourse), from the first dose of the study drug through 3 months after the last dose of the study drug. If the subject is routinely abstinent, the subject may use this form of contraception, but should choose a reliable form of contraception as mentioned above when the subject is no longer abstinent. Male subjects must not donate sperm from the first dose of the study drug until 3 months after the last dose.

Exclusion Criteria:

1. Be diagnosed with non-stable psoriasis or non-plaque psoriasis.
2. Presence of other inflammatory skin conditions in the treatment site that may confound the investigator's assessment of psoriasis.
3. Presence of significant pigmentary changes, scarring, sunburn, and other skin abnormalities in the treatment site that affect the assessment of psoriasis efficacy.
4. The treatment site is expected to be excessively exposed to natural/artificial light, tanning beds, or other LEDs within 4 weeks before the baseline visit and throughout the study.
5. Known hypersensitivity to any component of the test product or control product.
6. Current or prior hypercalcemia, vitamin D toxicity, severe renal insufficiency (Creatinine clearance <30 mL/min using the Cockcroft-Gault formula), or severe hepatic impairment (according to Child-Pugh C classification).
7. Systemic treatment with biological therapies.
8. Use of systemic agents for the treatment of psoriasis or any other agents which may influence the efficacy assessment of psoriasis within 4 weeks before the baseline visit or planned use during the study.
9. Use of psoralen plus ultraviolet A (PUVA) or ultraviolet B (UVB) phototherapy within 4 weeks before the first dose of this study or planned use during the study.
10. Use of topical medications for the treatment of psoriasis or any other agents which may influence the efficacy assessment of psoriasis within 2 weeks before the baseline visit.
11. Clinical signs of skin infection with bacteria, viruses, or fungi
12. Known Human Immunodeficiency Virus (HIV) infection, or hepatitis B, or hepatitis C, or syphilis.
13. Any chronic or acute medical condition that may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial.
14. Planned initiation or change in the use of an existing treatment that, in the opinion of the investigator, can affect the assessment of psoriasis efficacy.
15. Current participation in any other interventional clinical trial; or previous participation in a pharmaceutical clinical trial within 3 months or 5 half-lives (whichever is longer) or any other interventional clinical trial within 3 months prior to the first dose of this study.
16. Women who are pregnant, lactating, or planning to become pregnant during the study.
17. Major surgery within 4 weeks before the baseline visit or planned major surgery during the study.
18. Active infection requiring the application of oral or intravenous antibiotics, antifungals, or antivirals within 7 days before the baseline visit.
19. Cancer within 5 years before the first dose of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) success rate on the body (trunk and/or limbs) after 8 weeks of treatment with MC2-01 cream compared to vehicle and CAL/BDP gel in subjects with plaque psoriasis | Baseline and 8-week
  Proportion of subjects who achieve PGA treatment success (defined as a score of 0 or 1 plus a minimum 2-point decrease in PGA score from baseline) on the body (trunk and/or limbs) compared to after 8 weeks of treatment
  Psoriasis treatment success rate is measured at week 8 by the use of a Physician Global Assessment (PGA) score. Success is defined as a decrease from Baseline of minimum 2 point on a scale from 0 - 4, where: 0 = Clear; 1 = Almost clear; 2 = Mild Plaque thickening; 3 = Moderate Plaque thickening, 4 = Severe Plaque thickening.

SECONDARY OUTCOMES:
Percent change from baseline in mPASI after 8 weeks of treatment | Baseline and 8-week
  To evaluate the improvement in Modified Psoriasis Area and Severity Index (mPASI) after 8 weeks of treatment with MC2-01 cream compared to vehicle and CAL/BDP gel in subjects with plaque psoriasis.
  The extent and severity of the participant's psoriasis is assessed using a modified PASI scoring system (minus scalp, face, and flexures) at each 3 areas (arms, trunk and legs) using a scale from 0 - 6, where 0 = no psoriasis involvement and 6 = 90-100% involvement.
Assessment of Psoriasis Treatment Convenience Scale (PTCS) at week 8 of treatment | 8-week
  Subject assessment of treatment convenience using a Psoriasis Treatment Convenience Scale is defined as a sum of questions 1-5, where each question is scored on a scale from 1-10.
  How easy was the treatment to apply to the skin? "Very difficult" is 1 and "Very easy" is 10 How greasy was the treatment when applying it to the skin? "Very greasy" is 1 and "Not greasy" is 10 How moisturised did your skin feel after applying the treatment? "Not moisturized" is 1 and "Very moisturized" is 10 How greasy did your skin feel after applying the treatment? "Very greasy" is 1 and "Not greasy" is 10 How much did treating your skin disrupt your daily routine? "Very disturbing" is 1 and "Not disturbing" is 10.
PGA success rate on the scalp psoriasis after 8 weeks of treatment with MC2-01 cream compared to vehicle and CAL/BDP gel in subjects with plaque psoriasis | Baseline and 8-week
  Proportion of subjects with scalp psoriasis involved, PGA ≥2 and ≥0.3% body surface area (BSA) at baseline who achieve PGA treatment success on the scalp psoriasis after 8 weeks of treatment
Safety with MC2-01 cream in subjects with plaque psoriasis | 8-week
  Number of participants with adverse events and serious adverse events will be assessed.
Incidence of local skin reactions | 8 week
  Number of subjects that experience an local skin reactions by investigator assessment and local skin reactions reported as adverse events will be assessed
Number of Participants With Abnormal Electrocardiogram (ECG) Findings | 8 week
  Single measurements of 12-lead ECGs were obtained at Baseline to week 8, at any visit post-screen using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc).
Number of Participants With Vital Signs of Potential Clinical Importance | 8 week
  Body Temperature, Respiration, Pulse, and Blood Pressure were collected from participants for evaluation of vital signs by Potential Clinical Importance Criteria from Baseline to Week 8, any visit post-screen.

CONTACTS AND LOCATIONS:
Locations (55):
- China (55):
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Aerospace General Hospital, Beijing, Beijing Municipality
  - Bejjing Friendship Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Xiamen medical college, Xiamen, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Dermatology Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Third Affiliated Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Nanshan District People's Hospital, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Haikou Fifth People's Hospital, Haikou, Hainan
  - Chengde Medical University Affiliated Hospital, Chengde, Hebei
  - First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan University of Science and Technology Second Affiliated Hospital, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Taihe Hospital, Shiyan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan University of Medicine General Hospital, Huaihua, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital Of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng NO.1 People's Hospital, Yancheng, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shenyang Medical College Affiliated Central Hospital, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Jining NO.1 People's Hospital, Jining, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Chengdu Second People 's Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The First Affiliated Hospital of NingBo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No